CLINICAL TRIAL: NCT03156556
Title: Improving Access to Treatment of Anxiety and Depression in Young Adults Using Transdignostic iCBT: Feasibility of a Translated Version of an Empirically Supported Program
Brief Title: Improving Access to the Treatment of Anxiety and Depression Among Young Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universite de Moncton (Other)
Collaborators: Royal Bank of Canada (Unknown); MindCare Inc. (Unknown); Macquarie University, Australia (Other); University of Regina (Other); Horizon Health Network (Other)
Responsible Party: Principal Investigator, France Talbot, Associate professor, Universite de Moncton
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1617070
Record Dates: First submitted 2017-05-11; First posted 2017-05-17 (Actual); Last update posted 2022-06-02 (Actual); Status verified 2022-05

CONDITIONS: Generalized Anxiety Disorder; Major Depressive Disorder; Social Anxiety Disorder; Panic Disorder; Agoraphobia
MeSH Terms: conditions — Generalized Anxiety Disorder; Depressive Disorder, Major; Phobia, Social; Panic Disorder; Agoraphobia

STUDY DESIGN:
Intervention Model Description: 8-week pretest/post-test open trial including a 3-month follow-up.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mood Mechanic (Experimental): The Mood Mechanic Course is comprised of five online lessons completed over an 8-week period.
  * Lesson 1 presents information on anxiety and depression as well as on the cycle of symptoms.
  * Lesson 2 presents different strategies to generate helpful cognitions.
  * Lesson 3 describes strategies for physical de-arousal and for re-engaging in reinforcing activities.
  * Lesson 4 describes avoidance and safety behaviors and graded exposure.
  * Lesson 5 is about problem solving and relapse prevention.
  For each lesson, a "Do It Yourself" guide is included containing homework as well as case stories. Additional material on different topics is also included such as structured problem solving.
  Interventions: Behavioral: Mood Mechanic Course

INTERVENTIONS:
Behavioral: Mood Mechanic Course — French-Canadian version of the Mood Mechanic Course. Performed by a professional translator (Bourret Translation Inc.) and reviewed by the research supervisor, Professor France Talbot, clinical psychologist as well with expertise in CBT.
  Other Names: Cours Mécanique de l'Humeur (French-Canadian translation)

SUMMARY:
Anxiety and depression represent the most common mental health problems. Unfortunately, only a minority of people in need will seek or access traditional mental health services. Access to traditional psychological care is even more challenging for linguistic minorities as well as for people living in rural areas and for young adults - a group that has the highest rate of anxiety and depression but the lowest rate of consulting traditional services.Telepsychotherapy can facilitate access to effective psychological care as done in Australia where the government has been offering an evidence-based 8-week online therapy program called the Wellbeing Course. This online course helps people manage worry, stress, anxiety and depression. It has been evaluated in several clinical trials and successfully implemented as an Australian national treatment service. Its transdiagnostic nature, and the fact that the guidance of a clinician is not required for an efficient and safe administration and maintenance of therapeutic gains make it not only a viable option, but also an easily accessible fist line intervention. More recently, findings from a feasibility study conducted by our research laboratory have supported the efficacy of a French-Canadian translation among French-speaking minorities in New-Brunswick. A version of the Wellbeing Course for young adults has been developed called the Mood Mechanic Course. Empirical support has been obtained.

This study is a feasibility open trial, the first phase of a 3-phase research program designed to implement a French-Canadian translation of the Mood Mechanic Course in New Brunswick targeting groups for which access to traditional services has been most problematic: youth (18 to 25 years old), people living in rural areas and linguistic minorities. The course is an 8-week week program based on principles of cognitive behaviour therapy. It includes five online lessons, do-it-yourself exercises, case stories, and additional resources on different topic such as sleep hygiene. Twenty young adults will be recruited across New Brunswick among French-Canadian minority communities. Self-report measures assessing anxiety and depression will be administered pre/post treatment and at a 3-month follow-up. It is expected that the course will help overcome barriers in help seeking to improve the mental health of our communities.

DETAILED DESCRIPTION:
BACKGROUND. Anxiety and depression are highly prevalent mental health problems and chronic conditions accounting for the highest proportion of mental disorders in Canada. Young adults aged 15 to 24 are particularly vulnerable, this age group having the highest prevalence rates reported during a 12-month period of anxiety (11.6%) and depression (7%) in Canada. Access to evidence-based psychological treatments for anxiety and depression has been limited and particularly problematic for linguistic minorities.

RATIONALE FOR PERFORMING THE STUDY. Self-administered internet-based cognitive-behavioural therapy (iCBT) is a first-line therapy that could better meet the needs of young adults. Not only could its delivery format provide increased access to French services in both urban and rural areas, but it could also help young adults to overcome many of the barriers reported by Canadians with unmet or partially met needs for counselling.

An established iCBT shown to be effective for the treatment of anxiety and depression is the Wellbeing program developed by Titov and colleagues. The Wellbeing Course presents a number of advantages. It is a transdiagnostic program that allows the treatment of both anxiety and depression, which makes it a cost-efficient treatment. More recent evidence suggests that no direct clinical contact is required for gains to be significant and maintained over a 12-month follow-up. A version of the Wellbeing Course for young adults has been developed called the Mood Mechanic Course. Data gathered so far support its efficacy.

The majority of iCBT programs are only available in English, despite the fact that their translation can be a highly cost-effective strategy. More recently, findings from a feasibility study have supported the efficacy of a French-Canadian translation of the Wellbeing Course among French-speaking minorities in New-Brunswick.

PRIMARY OBJECTIVES. To examine the feasibility and acceptability of a French-Canadian and self-guided version of the Mood Mechanic Course on anxiety and depression among young adults.

SECONDARY OBJECTIVES. To assess the impact of the course on more specific symptoms of anxiety, resilience and life satisfaction.

HYPOTHESES. It is expected that:

* Participants will demonstrate a significant improvement from pre- to post-treatment on primary outcome measures of anxiety and depression and secondary outcome measures of life satisfaction.
* These improvements will be maintained during a three-month follow-up.
* Participants will report a high level of satisfaction with the course. No specific hypothesis is formulated regarding the impact of the Mood Mechanic Course on resilience as this component of the study is exploratory.

SAMPLE: A sample of 20 young adults will be recruited in among the general population New Brunswick using advertisements in various media as well as through a secure study website administered by Accra Solutions Inc (www.etherapies.ca). A sample of 20 to 25 participants has been recommended for feasibility or pilot studies when the aim is to demonstrate the efficacy in a single group and when the effect sizes will probably be moderate or large.

INTERVENTION. The Mood Mechanic Course is comprised of 5 online lessons completed over an 8-week period. For each lesson, a "Do It Yourself" guide is included containing homework as well as case stories and additional material on different topics.

INVESTIGATION PLAN. Young adults interested in the project will apply online through the website after reading a description of the project and filling out online questionnaires evaluating the study inclusion and exclusion criteria. A consent form will be sent electronically to applicants meeting the eligibility criteria. Entering their email address and clicking "I accept" will be considered as informed consent. A copy of the consent form will be sent to the participants through an encrypted email account created for the purpose of the study. Additional measures will be completed online as part of the pretest.

Applicants not meeting the study criteria will be sent an email to thank them for their interest in the study and will be provided a list of mental health resources. Applicants showing severe depression or suicidal thoughts will be encouraged to contact their family physician and will be sent a list of mental health resources as well.

Within one statutory day, candidates meeting the study criteria will receive an email informing them of their eligibility. Within five statutory days, participants will be contacted by phone to review the study procedures and to answer any questions that they may have. They will then be asked to provide contact information (i.e., name and phone number) and an emergency contact (either their family physician or a family member or friend) to be used only in the event that their state would significantly deteriorate. The outcome measures will be administered online through the secure study website using the software Ninja Forms.The lessons will be accessible through the secure study website using the Moodle software.

STANDARDIZED EMAILS. No contact with a clinician will be provided, but weekly contact will be maintained with the participants through standardized emails offering instructions, reminders and support.

SAFETY STUDY PROCEDURES. We are committed to the participants' safety. Safety measures will be included at all stages of this study based on Titov's procedures.

Screening and Selection: Just before applying to the study, it will be mentioned on the study website that this research project does not offer crisis or emergency services. Emergency contacts will be provided on the website.

During the study: All applicants will be informed (verbally and in writing) about the steps to take if they were to feel more distressed during the study, including contact details of the researchers, the importance of contacting their family physician, and contact details of emergency services. Applicants must also provide an emergency contact, be it their family physician or a family or friend who we will contact if we are concerned about the immediate state and safety of the participant (this is explained to the participants verbally, and in the Consent Form).

All participants' mood and symptoms will be monitored at the beginning of each new lesson using the Generalized Anxiety Disorder 7 item-scale (GAD-7) and Patient Health Questionnaire-9 items (PHQ-9). If participants' scores increase by more than 5 points from the pre-test and if the total score is ≥ 15 on the PHQ-9, they will receive an email including resources that can be used in case of an emergency. If participants' scores at the PHQ-9 is ≥ 23 or if they answer "3" on question 9 (suicidal ideation), the research director will contact them on the same day that the score is received to assess their situation and provide management. All adverse events will be promptly reported to the ethics committee of the Université de Moncton.

A list of mental health resources will be offered to all participants who will chose to end their participation during the study as well as at the end of the study. If participants withdrawing from the study present, based on their questionnaires, a deterioration of their state as described above, the same procedure will be followed.

At the 3-month follow-up, participants whose scores on the questionnaires indicate a clinical level of depression (>15 on the PHQ-9) or anxiety (> 10 on the GAD-7), will receive an email mentioning that if they wish to discuss their symptoms or other treatment options, we invite them to communicate with the research coordinator, or to indicate when it would be a good time for her to contact them. Otherwise we will encourage participants to communicate with their family physician or the closest mental health center to receive the necessary help, if it has not already been done. A mental health resource list will also be provided. If the scores indicate a severe level of depression (≥ 23 on the PHQ-9 or if they answer "3" on question 9), the same procedure as the one described above if such a situation were to happen during treatment, will be followed.

STATISTICAL ANALYSIS AND CLINICAL SIGNIFICANCE OF THE RESULTS. Changes in outcomes and maintenance of therapy gains will be evaluated using one-way repeated measures ANOVAs. Missing data will be handled using the last observation carried forward (LOCF). Two indices of clinical improvement will be estimated: remission and recovery rates.

DATA SAFETY. All data collected as part of this research will remain confidential except in the case of a breach of confidentiality if a participant presented, for example, an immediate risk of harm. Participants must create a username and password that will be used to complete the online questionnaires. Standardized emails will be sent to participants from a encrypted email account created by Accra Solutions Inc. for the purposes of the study. Only the name of the participants will be included in these emails, to which they will have consented. To maintain participants' privacy and confidentiality, they will not be able to use a username that contains identifiable information (e.g., real name, address, city you live in). They will be asked to create a username of four letter (four first letters of their mother or father's name) and four numbers (day and month of their birthday). The participants will generate a password. It will be specified to use a secure one made of 8 characters including letters, numbers and a special character.Only researchers of the study, the system administrator and Macquarie University will have access to the data as specified in the consent form and as specified in the memorandum of understanding with Macquarie University.

STORAGE AND ARCHIVING OF STUDY DOCUMENTS. The consent form and the identification form including the contact information and password will be printed and kept in a locked filing cabinet in the office of Professor France Talbot, research director. All electronic data will be stored in a secure database within https://www.etherapies.ca. A data file will be created in SPSS for all data and will be stored on a computer in the research director's research laboratory, the Telepsychotherapy Unit. The names of the participants will not appear in this file, only their password. As well, a password is required to access the files on this computer. The data file will be saved on a USB key kept in a locked filing cabinet in the Telepsychotherapy Unit. The information gathered during the study will be destroyed after 5 years. The data file will be kept seven years following the publication of the results, and then destroyed.

ELIGIBILITY:
Inclusion Criteria:

* Resident of New Brunswick;
* 18 to 25 years of age;
* French as their native language;
* Good comprehension of written French;
* Reliable access to the Internet;
* Clinical levels of depression, generalized anxiety disorder, panic disorder or social anxiety disorder, as indicated by the total score of at least one of the following measures: QSP-9 ≥ 5; GAD-7 ≥ 5, PAS ≥ 19, SPIN ≥ 19;
* Not currently following another cognitive-behavioral therapy (CBT);
* No change of medication at least one month prior to the study and no change expected over the next two months;
* In agreement to share relevant personal information.

Exclusion Criteria:

* Severe depression or suicide intent or plan (score ≥ 23 or a score > 2 on item 9 (suicidal ideation) of PHQ-9;
* Currently experiencing psychotic symptoms.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2017-05-15 (Actual); Primary Completion 2018-01-31 (Actual); Study Completion 2018-01-31 (Actual)

PRIMARY OUTCOMES:
Changes in depression as assessed with the Patient Health Questionnaire-9 items | Pre-test (Week 1), Post-test (Week 8) and 3-month follow-up
  French version: 9 items assessing symptoms of major depressive disorder on a scale from 0 (Not at all) to 3 (Nearly every day).
Changes in anxiety as assessed with the Generalized Anxiety Disorder Scale 7-Item Scale | Pre-test (Week 1), Post-test (Week 8) and 3 month follow-up
  French version: 7 items assessing symptoms of generalized anxiety disorder on a scale from 0 (Not at all) to 3 (Nearly every day).

SECONDARY OUTCOMES:
Changes in anxiety as assessed with the Panic and Agoraphobia Scale (PAS) | Pre-test (Week 1), Post-test (Week 8) and 3 month follow-up
  French version: 14 items assessing symptoms of panic attacks, panic disorder and agoraphobia.
Changes in anxiety as assessed with the Social Phobia Inventory (SPIN) | Pre-test (Week 1), Post-test (Week 8) and 3 month follow-up
  French version: 17 items assessing symptoms of social anxiety disorder on a scale from 0 (Not at all) to 4 (Extremely).
Changes in resilience as assessed with the Connor-Davidson Resilience Scale | Pre-test (Week 1), Post-test (Week 8) and 3 month follow-up
  French version: 25 items assessing psychological resilience on a scale from 0 (Not at all true) to 4 (True nearly all the time).
Changes in life satisfaction as assessed with the Life Satisfaction Questionnaire | Pre-test (Week 1), Post-test (Week 8) and 3 month follow-up
  French version: 5 items assessing life satisfaction using a scale from 1 (Strongly disagree) to 7 (Strongly agree).
Treatment acceptability | Post-test (Week 8)
  Four questions: (1) 'Overall, how satisfied were you with the Course?', (2) 'How satisfied were you with the Lessons and Lesson Summaries?', (3) 'Would you feel confident in recommending this treatment to a friend?', and (4) 'Was it worth your time doing the Course?' These questions have been used in previous research examining the acceptability of iCBT (e.g., Titov et al., 2013). For the purposes of revising and improving the program for future studies among Francophone minority communities, participants will also be asked to provide feedback about the program over the phone at post-treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Josée LeBlanc, B.A., Principal Investigator — Université de Moncton; France Talbot, Ph.D., Study Director — Université de Moncton
Locations (1):
- Université de Moncton, Moncton, New Brunswick, Canada

IPD SHARING:
Plan to Share IPD: No